CLINICAL TRIAL: NCT06726369
Title: A Phase 1 Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of MK-6204 (SKB535) for Injection in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-6204-001/SKB535-I-01
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
Keywords: ADC; safety; tolerability; pharmacokinetics
MeSH Terms: interventions — WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MK-6204 (SKB535) for Injection (Experimental): Several dose levels of MK-6204 (SKB535) for Injection are planned and administered every 3 weeks.
  Interventions: Drug: MK-6204 (SKB535) for Injection

INTERVENTIONS:
Drug: MK-6204 (SKB535) for Injection — MK-6204 (SKB535) for injection is administered every 3 weeks (q3w) until radiographic disease progression (PD), intolerable toxicity, death, or discontinuation of treatment, whichever occurs first.

SUMMARY:
This is an open-label, nonrandomized, multicenter, Phase 1 study to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of MK-6204 as monotherapy in participants with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, nonrandomized, multicenter, Phase 1 study to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of MK-6204 as monotherapy in participants with advanced solid tumors. The primary objectives are to evaluate the safety and tolerability of MK-6204. The secondary endpoints include PK parameters, ORR, DOR, and immunogenicity of MK-6204. The study will include a Screening Phase, a Treatment Phase, and a Post-treatment Follow up Phase.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Have a histologically or cytologically confirmed advanced/metastatic solid tumor by pathology report and have failed or do not have available standard treatments. The tumor types will be limited to: CRC; Gastric carcinoma or gastroesophageal junction (GEJ) adenocarcinoma; Esophageal carcinoma; Pancreatic cancer; NSCLC; Cervical carcinoma; Head and Neck squamous cell carcinoma.
3. Have measurable disease by RECIST 1.1 as assessed by the local site investigator/radiology. Target lesions situated in a previously irradiated area are considered measurable if progression has been shown in such lesions.
4. Have a performance status of 0 or 1 on the ECOG Performance Scale.
5. The participant has provided documented informed consent for the study.
6. Participants who agree to provide archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated.
7. Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible.

Exclusion Criteria:

1. Active severe digestive disease, including but not limited to complete or incomplete gastric outlet obstruction, persistent/recurrent vomiting, severe gastrointestinal hemorrhage, gastric or duodenal ulcers, acute gastrointestinal perforation, acute necrotizing pancreatitis, ulcerative enteritis, congenital megacolon, or Crohn's disease.
2. Participants with a history of interstitial lung disease (ILD) or a history of noninfectious pneumonitis that required steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
3. Received strong cytochrome P450 (CYP3A4) inhibitors or inducers within 2 weeks prior to the first dose of study intervention or within 5 half-lives of drug elimination, whichever is longer.
4. Received strong breast cancer resistance protein (BCRP) inhibitors within 2 weeks prior to the first dose of study intervention or within 5 half-lives of drug elimination, whichever is longer.
5. Received prior systemic anticancer therapy including investigational agents within 4 weeks or 5 half-lives, whichever is shorter, before intervention allocation.
6. Known additional malignancy that is progressing or has required active treatment within the past 2 years.
7. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable (i.e., without evidence of progression) for at least 4 weeks as confirmed by repeat imaging performed during the study screening, are clinically stable and have not required steroid treatment for at least 14 days before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | From the date of first dose until up to 21 days of intervention
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during the evaluation period and is at least possibly related to study drug.
Adverse Event (AE) | From the date of first dose until up to 30 days after the last dose of intervention
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention.
Serious Adverse Event (SAE) | From the date of first dose until up to 30 days after the last dose of intervention
  An SAE is defined as any serious untoward medical occurrence that meets the pre-specified criteria in the protocol

SECONDARY OUTCOMES:
PK parameter AUC | Through study completion, an average of 2 years
  PK parameter AUC after single and multiple doses
PK parameter Cmax | Through study completion, an average of 2 years
  PK parameter Cmax after single and multiple doses
PK parameter Cmin | Through study completion, an average of 2 years
  PK parameter Cmin after single and multiple doses
Objective response rate (ORR) | Through study completion, an average of 2 years
  ORR refers to the proportion of participants who have achieved confirmed complete response (CR) or partial response (PR).
Duration of response (DOR) | Through study completion, an average of 2 years
  DOR refers to the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Immunogenicity of MK-6204 | Through study completion, an average of 2 years
  ADA incidence

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Shanghai East Hospital, Shanghai
  - Hubei Cancer Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: No